CLINICAL TRIAL: NCT04651491
Title: Study of Antiviral Therapy of Influenza and ARVI With Kagocel ® in Children
Brief Title: Treatment of Influenza and ARVI in Children by Kagocel ®
Status: Completed | Type: Observational
Sponsor: Nearmedic Plus LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: version 2.0 from 10.02.2015
Record Dates: First submitted 2020-11-23; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2016-09

CONDITIONS: Influenza; Acute Upper Respiratory Infection
Keywords: influenza; flu; acute respiratory viral infection; ARVI; acute upper respiratory infection; AURI
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Therapy with interferons' inducers: Therapy according to routine practice (including Kagocel)
  Interventions: Drug: Kagocel

INTERVENTIONS:
Drug: Kagocel — The researchers prescribed antiviral medications, including Kagocel, according to routine clinical practice. Patients who were assigned Kagocel were invited to participate in the study.
  Kagocel administration:
  1. for children from 3 to 6 years old (n=41): In the first 2 days - 1 tablet 2 times a day, in the next 2 days - 1 tablet once a day. Total for the course of administration 6 tablets within the period of 4 days.
  2. for children from 6 years old (n=39) - administered in the first 2 days - 1 tablet 3 times a day, in the next 2 days - 1 tablet 2 times a day. Total for the course of administration 10 tablets within the period of 4 days.

SUMMARY:
This study examined the etiology of acute respiratory viral infections (ARVI) during the 2015-2016 season, evaluated the statistics of the incidence of influenza and ARVI in this period (epidemiology: severity of the disease and bacterial exacerbations; demographics of patients; duration and timing of treatment; safety; quality of treatment), and evaluated the effectiveness of complex therapy with an emphasis on the using of interferon inducers in hospitalized children aged 3 to 11 years.

DETAILED DESCRIPTION:
This non-interventional observational study included 80 patients aged 3 to 11 years who were hospitalized with influenza and acute respiratory viral infections (ARVI) symptoms at any time from the onset of the disease (up to 15 days) and who were prescribed the interferon inducer Kagocel as an antiviral medicine.

The diagnosis of influenza and ARVI was confirmed in accordance with the world health organization (who) guidelines for the pharmacological treatment of pandemic influenza A (H1N1) 2009 and other influenza viruses.

All patient examinations are conducted in accordance with local routine clinical practice and local and international standards of care.

After the end of treatment, the following data were collected and analyzed:

* demography
* disease severity
* anamnesis data (data of influenza vaccination in the current season; pre-school facilities visits; previous contacts with a patient with influenza / ARVI; previous antiviral therapy for the current episode of the disease; concomitant diseases)
* body temperature (morning/evening)
* chills and fever (cumulative score based on all symptoms: 0-no symptoms, 1-mild, 2-moderate, 3-severe)
* intoxication symptom (cumulative score based on all symptoms: 0-no symptoms, 1-mild, 2-moderate, 3-severe)
* catarrhal symptoms (cumulative score based on all symptoms: 0 - no symptoms, 1-mild, 2-moderate, 3-severe)
* timelines: the beginning of the disease, the first visit to the doctor, the beginning of treatment, the duration of the disease
* determination the causative agent by PCR (on presentation of patients and their discharge on 5-6 days from start of therapy)
* antiviral therapy (Kagocel dose depending on age)
* symptomatic treatment of the current episode of influenza or ARVI before and during the patient's hospitalization
* bacterial exacerbations (Yes/no)
* treatment of bacterial exacerbations (drug name)
* adverse events

ELIGIBILITY:
Inclusion Criteria:

1. The patient's age from 3 to 11 years inclusive.
2. The patient was hospitalized with symptoms of influenza and ARVI.
3. The appointment of drug Kagocel ® as an antiviral therapy of influenza or ARVI by the doctor during hospitalization
4. No history of allergy and / or hypersensitivity to the components of the drug Kagocel ® .
5. Signed informed consent to participate in the study.

Exclusion Criteria:

- patients who received antiviral and immunomodulatory medications within 15 days prior to hospitalization

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients with confirmed diagnosis of influenza or influenza-like illness caused by a different type of virus which are on anti-flu therapy
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-09-11 (Actual); Primary Completion 2016-05-05 (Actual); Study Completion 2016-09-28 (Actual)

PRIMARY OUTCOMES:
Changes in the number of respiratory viruses in nasopharyngeal smears by multiplex PCR | 2 points: day of hospitalization and 5-6 day of treatment
  Identification of respiratory viruses such as influenza a and b, human respiratory syncytial virus, parainfluenza viruses of types 1-4, coronaviruses, metapneumoviruses, rhinoviruses, adenoviruses of groups B, C, E, and bokaviruses, and assessment of the duration of their isolation
Duration and severity of fever in patients with influenza and in patients with ARVI | up to 7 days (at least)
The dynamics and the severity of intoxication and catarrhal syndromes in patients with influenza and in patients with ARVI | up to 7 days (at least)
  Intoxication syndrome: drowsiness, muscle pain, weakness, sweating, chills, eye pain, headache.
  Catarrhal syndromes: pharyngeal hyperemia, cough, rhinorrhea, nasal congestion, sore throa.
  Qualitative signs were evaluated in points-absence of a sign-0 points, weakly expressed sign - 1 point, medium (moderate) expressed-2 points, bright (strongly) expressed-3 points
Number of participants with symptoms of ARVI or influenza | up to 7 days (at least)
  Number of patients with intoxication syndrome (drowsiness, muscle pain, weakness, sweating, chills, eye pain, headache), catarrhal syndromes (pharyngeal hyperemia, cough, rhinorrhea, nasal congestion, sore throa) and fever
Number of participants who required antibiotic therapy | up to 7 days (at least)
Number of participants with ARVI and influenza complications | up to 7 days (at least)

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events (AE) with regards to type and severity of AE (mild, moderate, severe; according to physician's opinion) | up to 7 days (at least)

CONTACTS AND LOCATIONS:
Overall Officials: Irina Babachenko, Professor, Dr. habilitated, Principal Investigator — Research Institute of Children's Infections of the Federal Medical and Biological Agency,
Locations (1):
- Research Institute of Children's Infections of the Federal Medical and Biological Agency,, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sharipova E.V., Babachenko I.V., Levina A.S., Grigoriev S.G. Antiviral therapy of acute respiratory viral infection and influenza in children in a hospital. Journal Infectology. 2018;10(4):82-88. (In Russ.) doi.org/10.22625/2072-6732-2018-10-4-82-88 — http://journal.niidi.ru/jofin/article/view/808
- See also: Babachenko I.V., Sharipova E.V., Belikova T.L. Hospital- and clinic-based approaches to the treatment of ARVI in children. Meditsinskiy sovet = Medical Council. 2017;(1):94-99. (In Russ.) https://doi.org/10.21518/2079-701X-2017-1-94-99 — https://med-sovet.pro/jour/article/view/1684